CLINICAL TRIAL: NCT06139614
Title: Personal Resilience Skills to Improve Surgery Training (PERSIST)
Brief Title: Personal Resilience Skills to Improve Surgery Training
Acronym: PERSIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00113779
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Well-Being, Psychological; Anxiety Depression
Keywords: Personal resilience; Professional Fulfillment; Positive Well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: There will be one group of Junior Assistant Residents (JAR, N = 10) and one group of Senior Assistant Residents (SAR, N =10), which will be conducted separately. At baseline, all participants will complete questionnaires related personal resilience, including professional fulfillment (professional fulfillment, work exhaustion, interpersonal disengagement), depression symptoms, anxiety, symptoms, self-valuation, flourishing, and psychosocial working conditions. At post-treatment (end of session 8), participants will complete the baseline questionnaires (with the exception of psychosocial working conditions), as well as a questionnaire assessing acceptability of the group experience and content. The post-treatment questionnaires will be repeated as a 3-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assistant Residents (Experimental): At baseline, all participants will complete questionnaires related personal resilience, including professional fulfillment (professional fulfillment, work exhaustion, interpersonal disengagement), depression symptoms, anxiety, symptoms, self-valuation, flourishing, and psychosocial working conditions. At post-treatment (end of session 8), participants will complete the baseline questionnaires (with the exception of psychosocial working conditions), as well as a questionnaire assessing acceptability of the group experience and content. The post-treatment questionnaires will be repeated as a 3-month follow-up.
  Interventions: Behavioral: PERSIST

INTERVENTIONS:
Behavioral: PERSIST — PERSIST is adapted from empirically validated treatment of negative affect and low positive emotion. Skills Training 1 includes content across 4 sessions on 1) understanding emotions, 2) present-moment emotional awareness, 3) cognitive flexibility, and 4) countering avoidant and emotion-driven responses. Skills Training 2 includes content across 4 sessions on a) translating values to action, b) lower barriers to action, c) countering avoidance, and d) maintaining actions that support personal resilience. The classes will occur every other Wednesday, resulting in a 16-week intervention period.

SUMMARY:
The objective of the current study (PERSIST) is to 1) determine acceptability of an 8-session (16 week) group curriculum on personal resilience skills for residents in the Duke General Surgery Program, and 2) examine changes in professional fulfillment, depression symptomatology, anxiety symptomatology, and self-valuation, and positive wellbeing (flourishing) at the end of the program and 3-month follow-up compared to baseline, 3) examine performance on surgery training metrics compared to the mean performance of non-participants. Participants will be residents active in the Duke General Surgery Program. There will be one group of Junior Assistant Residents (JAR, N = 10) and one group of Senior Assistant Residents (SAR, N =10), which will be conducted separately. At baseline, all participants will complete questionnaires related personal resilience, including professional fulfillment (professional fulfillment, work exhaustion, interpersonal disengagement), depression symptoms, anxiety, symptoms, self-valuation, flourishing, and psychosocial working conditions. At post-treatment (end of session 8), participants will complete the baseline questionnaires (with the exception of psychosocial working conditions), as well as a questionnaire assessing acceptability of the group experience and content. The post-treatment questionnaires will be repeated as a 3-month follow-up. All study activities are considered low risk, and there the training is expected to have the benefit of teaching lasting skills to promote professional and personal resilience. To protect participant confidentiality, surgery staff and faculty will not have access linkage between study variables and participant identity.

DETAILED DESCRIPTION:
The primary aims/objectives are to examine acceptability of the PERSIST intervention, and pre-post changes relevant to resident resilience, as operationalized in measures of personal and professional well-being. The investigators intend to enroll both Junior Assistant Residents (JAR) and Senior Assistant Residents (SAR) cohorts in a combined sample; and secondarily results by group.

The secondary objective is to examine whether participation in PERSIST is associated with better training and safety outcomes compared to resident who do not participate.

Aim 1: Determine acceptability of an 8-session PERSIST intervention for General Surgery residents.

Aim 2: Assess change on measures of personal and professional well-being following an 8 session PERSIST intervention for General Surgery residents. The investigators anticipate that individuals completing PERSIST will show improvement in professional fulfillment, depression symptoms, anxiety symptoms, flourishing, and self-valuation at post-treatment and 3-month follow up compared to baseline.

Aim 3: Compare training and safety outcomes of PERSIST participants compared to non-participants.

PERSIST is adapted from empirically validated treatment of negative affect and low positive emotion. Skills Training 1 includes content across 4 sessions on 1) understanding emotions, 2) present-moment emotional awareness, 3) cognitive flexibility, and 4) countering avoidant and emotion-driven responses. Skills Training 2 includes content across 4 sessions on a) translating values to action, b) lower barriers to action, c) countering avoidance, and d) maintaining actions that support personal resilience. The classes will occur every other Wednesday, resulting in a 16-week intervention period.

The investigators plan to collect multiple sources of information on acceptability. Primarily this will be via questionnaire rating of the experience and value of the 8 content topics in PERSIST. Additionally, the investigators will review and categorize response from open ended content, track participant attendance over the duration of the intervention, and document any feasibility issues related to recruitment, attendance, or dissemination of content. All measures related to well-being assessed at pre-intervention, post-intervention, and 3-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* The pilot cohort will be composed of junior assistant residents (JAR) and senior assistant residents (SAR) members of the Duke General Surgery Residency Program.

Exclusion Criteria:

* Because the PERSIST intervention is focused on coaching resilience to the challenges of clinical training, JAR and SAR who will be completing a research year during the intervention period will be excluded from participation.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Program Acceptability as measured by participant attendance in mean percent | Intervention end - 16 weeks
  Investigators will track participant attendance over the duration of the intervention and report in total mean percent.
Program Acceptability as measured by Questionnaire | Intervention end - 16 weeks
  A questionnaire rating of the experience and value of the 8 content topics in PERSIST using a scale of 5-50 (higher score = higher acceptability).
Professional Well-being as measured by the Professional Fulfillment Index (PFI) | 3 months post-intervention
  Overall professional well-being will be assessed with the Professional Fulfillment Index (PFI), which is scored on a scale of 0-24 (higher score = better outcome).
Personal Well-being as measured by the Self-Valuation (S-V) scale | 3 months post-intervention
  Personal well-being will be assessed with the Self-Valuation scale (S-V), which is scored on a scale of 0-16 (higher score = better outcome).
Positive well-being as assessed by the Flourishing Scale (FS) | 3 months post-intervention
  Positive well-being will be assessed by the Flourishing Scale (FS), which is scored on a scale of 8-56 (higher score = better outcome).
Exhaustion as measured by the Professional Fulfillment Index (PFI) | 3 months post-intervention
  Exhaustion from work will be assessed with the Professional Fulfillment Index (PFI), which is scored on a scale of 0-44 (higher score = worse outcome).
Anxiety symptoms as measured by the General Anxiety Disorder-7 questionnaire (GAD-7) | 3 months post-intervention
  Anxiety symptoms will be assessed using the General Anxiety Disorder-7 questionnaire (GAD-7), which is scored on a scale from 0-21 (higher = worse outcome).
Depression symptoms as measured by the 8-item version of the Patient Health Questionnaire (PHQ-8) | 3 months post-intervention
  Depression symptoms will be assessed using the 8-item version of the Patient Health Questionnaire (PHQ-8), which is scored on a scale from 0-24 (higher = worse outcome).

SECONDARY OUTCOMES:
Clinical and professional competencies measured by milestone achievement in Entrustable Professional Activities (EPA) | 3 months post-intervention
  Clinical and professional competencies will be assessed by milestone achievement in Entrustable Professional Activities (EPA). EPA scores are core metrics for evaluating resident performance and providing feedback within the General Surgery Program.
  Surgery training outcomes occur in the normal course of training and are not expressly collected as part of the PERSIST intervention. ABSITE and EPA scores are core metrics for evaluating resident performance and providing feedback within the General Surgery Program.
Safety outcomes as measured by mean number of Safety Reporting System (SRS) incidents | 3 months post-intervention
  Safety outcomes will be assessed by mean number of Safety Reporting System (SRS) incidents compared to non-participants.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Tracy, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No